CLINICAL TRIAL: NCT07182344
Title: Effects of iTBS on Cognitive Control in Children With ADHD: A Randomized, Sham-Controlled Study Integrating EEG During ANT, fNIRS, MRI, and Genetic Markers
Brief Title: Brain Stimulation and Attention Control in Children With ADHD
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Neurolab Plus (Industry)
Collaborators: Al-Farabi Kazakh National University (KazNU) (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2.2.6.2; BR27198099 (Other Grant/Funding Number: Non-profit joint-stock company "Al-Farabi Kazakh National University")
Record Dates: First submitted 2025-08-20; First posted 2025-09-19 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-08

CONDITIONS: ADHD - Attention Deficit Disorder With Hyperactivity
Keywords: Transcranial Magnetic Stimulation; Theta Burst Stimulation; Pediatric Neurostimulation; Neurodevelopmental Disorders; Multimodal Biomarkers; Electrophysiology; Functional Near-Infrared Spectroscopy; Magnetic Resonance Imaging; Genetic Markers; Randomized Controlled Trial; Sham-Controlled Trial; Child Neuropsychology; Attention Deficit Disorder with Hyperactivity; Executive Function; Cognitive Control; Attention Network Test; Prefrontal Cortex Excitability
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity; Neurodevelopmental Disorders

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Participants, care providers, investigators, and outcome assessors are all blinded to group assignment (active vs. sham TMS). The sham condition mimics the sound and sensation of stimulation without delivering active magnetic pulses, using an identical setup. Randomization and group codes are maintained by an independent administrator and not revealed until after final data analysis. Blinding is used to reduce bias in behavioral, neurophysiological, and questionnaire-based outcomes.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active iTBS to Right DLPFC (Experimental): Participants receive active intermittent theta burst stimulation (iTBS) to the right dorsolateral prefrontal cortex (DLPFC). Each session includes 600 pulses delivered in 2-second trains of 50 Hz bursts (triplets at 5 Hz), repeated every 10 seconds for a total duration of approximately 3 minutes, at 80% of active motor threshold. A total of 10 sessions is administered across two weeks.
  Interventions: Device: Intermittent Theta Burst Stimulation to Right DLPFC
- Sham iTBS (Right DLPFC) (Sham Comparator): Participants receive sham stimulation over the right DLPFC using the same coil orientation, session structure, and auditory cues as the active iTBS group, but without magnetic field induction. Ten sham sessions are delivered over two weeks to maintain blinding and control for placebo effects.
  Interventions: Device: Sham Intermittent Theta Burst Stimulation

INTERVENTIONS:
Device: Intermittent Theta Burst Stimulation to Right DLPFC — Participants receive intermittent theta burst stimulation (iTBS) applied to the right dorsolateral prefrontal cortex (DLPFC). The protocol consists of 600 pulses delivered in bursts of 3 pulses at 50 Hz, repeated at 5 Hz for 2 seconds, every 10 seconds, over approximately 3 minutes per session. Stimulation is delivered at 80% of the participant's active motor threshold. Ten sessions are administered across two weeks.
  Other Names: iTBS
  Arms: Active iTBS to Right DLPFC
Device: Sham Intermittent Theta Burst Stimulation — Participants receive sham intermittent theta burst stimulation (iTBS) to the right dorsolateral prefrontal cortex (DLPFC) using a placebo coil. The coil replicates the sound and scalp sensation of active stimulation without generating sufficient magnetic output to alter cortical excitability. Session length, coil placement, and stimulation parameters are matched to the active iTBS condition. To preserve blinding, both participants and administering staff wear earplugs to minimize auditory differences between sham and active coils. This condition serves as a placebo control for evaluating iTBS effects on attention in children with ADHD.
  Other Names: Sham iTBS
  Arms: Sham iTBS (Right DLPFC)

SUMMARY:
The goal of this clinical trial is to learn if brain stimulation can help children ages 6 to 12 with attention-deficit/hyperactivity disorder (ADHD) improve their attention and self-control. The main questions it aims to answer are:

Does intermittent theta burst stimulation (iTBS) improve performance on a task that tests attention and reaction times? Can brain activity and genetics help predict who benefits most from this treatment?

Researchers will compare randomly assigned active iTBS to sham (inactive) stimulation groups to see if the treatment helps.

Participants will:

Receive 10 sessions of either active or sham iTBS over 2 weeks Complete a computer task measuring attention before and after stimulation Wear a brain cap during the task to record EEG signals, also take part in resting-state brain scans, namely magnetic resonance imaging (MRI) and functional near-infrared spectroscopy (fNIRS), and provide a saliva sample for genetic testing

DETAILED DESCRIPTION:
This study explores whether noninvasive brain stimulation can improve attention control in children diagnosed with Attention-Deficit/Hyperactivity Disorder (ADHD), and how biological factors such as brain activity, brain structure, and genetics may predict individual differences in response. The primary focus is on executive attention-the ability to focus on relevant information, ignore distractions, and resolve conflicts between competing signals. These skills are often impaired in children with ADHD and closely linked to underlying differences in brain function.

To address this, the study uses intermittent theta burst stimulation (iTBS), a specialized form of transcranial magnetic stimulation (TMS). This method delivers rapid bursts of magnetic energy in intervals that are designed to increase the excitability of the targeted brain region. The stimulation is applied to the right dorsolateral prefrontal cortex (DLPFC), a key area involved in attention regulation, response inhibition, and cognitive control-functions that are often altered in ADHD.

A total of 40 children between the ages of 6 and 12 will participate. All must have a confirmed diagnosis of ADHD, verified through structured clinical evaluation. To ensure task comprehension and protocol tolerance, all participants must meet a minimum cognitive ability threshold based on a brief IQ screening.

Participants are randomly assigned to receive either active iTBS or sham stimulation. In the sham condition, the procedures and equipment appear identical, but the stimulation coil is positioned in a way that does not affect brain activity. This ensures that results can be attributed to the stimulation itself rather than expectations or placebo effects. Both participants and researchers conducting assessments are unaware of group assignments to maintain blinding.

Each participant undergoes ten sessions of either active or sham iTBS, typically spaced across two weeks. The stimulation protocol is brief-each session lasting only a few minutes-and individualized according to motor threshold testing, which ensures the intensity is appropriate and safe for each child. All procedures are delivered under professional supervision in a child-friendly environment with appropriate hearing protection.

To assess attentional performance, children complete the Attention Network Test (ANT) before and after the stimulation phase. This computerized task measures three key domains of attention: alerting, orienting, and executive control. During the task, children respond to the direction of arrows on the screen, which may be surrounded by distracting cues. This allows researchers to calculate specific reaction-time profiles associated with attention and conflict resolution.

While the ANT is being performed, the study also records electroencephalographic (EEG) data to capture the brain's electrical responses to each trial. EEG is a noninvasive method that tracks fast neural signals in real time using a cap placed on the child's head. It allows for detailed analysis of how the brain prepares for, reacts to, and regulates attentional demands-especially in the milliseconds following stimulus presentation.

In addition, resting-state fNIRS recordings are collected before and after the intervention. fNIRS is a child-friendly brain imaging method that uses near-infrared light to measure blood oxygen levels in the cortex. When the child is at rest, this technique provides insight into the baseline functional state of the DLPFC, allowing researchers to detect changes in regional activation associated with the stimulation.

To explore whether structural brain features may predict stimulation outcomes, each participant also undergoes a one-time MRI scan. This provides high-resolution images of brain anatomy and can reveal differences in cortical thickness, brain volume, or regional structure that may relate to ADHD symptoms or treatment response.

Finally, the study collects genetic material from saliva samples to investigate specific single-nucleotide polymorphisms in genes linked to dopamine signaling, synaptic function, or neurodevelopment. These include candidate genes such as DRD4, DAT1, COMT, and SLC6A3, which have been associated with attentional control and ADHD phenotypes. Genetic data will be used to explore biological moderators of iTBS efficacy.

This multimodal approach-combining behavioral, electrophysiological, neuroimaging, and genetic methods-aims to move beyond the question of whether iTBS is effective for ADHD. Instead, it seeks to understand how and for whom it works, contributing to the long-term development of individualized, evidence-based neuromodulation strategies for children with attentional difficulties.

The study complies with ethical standards for pediatric research and brain stimulation, and is overseen by the Local Ethical Committee of Al-Farabi Kazakh National University. It is funded by the Ministry of Science and Higher Education of the Republic of Kazakhstan under grant number IRN BR27198099. No U.S. FDA-regulated products are involved.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 6-12 years at the time of enrollment.
* Clinical diagnosis of Attention-Deficit/Hyperactivity Disorder (ADHD), any presentation type, confirmed using the Vanderbilt ADHD Diagnostic Parent Rating Scale and clinical interview.
* Intelligence quotient (IQ) ≥ 70 as measured by the General Ability Index (GAI) from the Wechsler Intelligence Scale for Children - Fifth Edition (WISC-V).
* Ability to understand and follow instructions for the Attention Network Test (ANT) and stimulation procedure.
* Stable medication regimen for ADHD (if any) for at least 4 weeks before the start of the study.
* Written informed consent from a parent or legal guardian, and assent from the child when appropriate.

Exclusion Criteria:

* History of epilepsy, seizures, or abnormal EEG suggestive of seizure risk.
* Presence of metal implants, devices, or foreign bodies in or near the head (except dental fillings) that are contraindicated for TMS or MRI.
* Serious neurological disorders other than ADHD (e.g., cerebral palsy, brain injury, neurodegenerative disease).
* Severe psychiatric disorders requiring hospitalization or urgent intervention.
* Current or past history of significant head trauma with loss of consciousness > 5 minutes.
* Uncorrected hearing or vision problems that could interfere with task performance.

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Estimated)
Dates: Start 2025-09-04 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Change in Executive Attention Efficiency as Measured by the Attention Network Test (ANT) | Baseline and post-intervention (within 7 days of final TMS session)
  Executive attention is measured as the conflict effect (reaction time in incongruent flanker trials - reaction time in congruent flanker trials). Smaller values of reaction time difference (milliseconds, ms) reflect improved conflict resolution and executive control.

SECONDARY OUTCOMES:
Change in Event-Related Potentials During ANT (EEG - N2 Component) | Baseline and up to 7 days after the final TMS session.
  Amplitude of N2 (~200-350 ms) during ANT incongruent vs. congruent trials, reflecting conflict monitoring (µV²/Hz).
Change in Event-Related Potentials During ANT (EEG - P3 Component) | Baseline and up to 7 days after the final TMS session.
  Amplitude of P3 (~350-550 ms) during ANT trials, reflecting attentional allocation (µV²/Hz).
Change in Oscillatory EEG Power During ANT (Theta Band) | Baseline and up to 7 days after the final TMS session.
  Mean theta-band power (4-7 Hz) over fronto-central electrodes during ANT (µV²/Hz).
Change in Resting-State Prefrontal Activity - Mean Oxygenation (fNIRS) | Baseline and up to 7 days after the final TMS session.
  Resting-state functional near-infrared spectroscopy (fNIRS) measurement of mean oxygenated hemoglobin (HbO, µM) in the dorsolateral prefrontal cortex (DLPFC).
Change in Resting-State Prefrontal Activity - Functional Connectivity (fNIRS) | Baseline and up to 7 days after the final TMS session.
  Resting-state fNIRS measurement of connectivity indices across DLPFC channels (e.g., correlation coefficients between HbO time series).
Change in ADHD Symptom Severity (Vanderbilt ADHD Diagnostic Parent Rating Scale, VADPRS) | Baseline and up to 7 days after the final TMS session.
  Parent-reported Vanderbilt ADHD Diagnostic Parent Rating Scale (VADPRS). The questionnaire includes 47 symptom items scored 0-3 ("Never" to "Very Often"), covering inattention, hyperactivity/impulsivity, oppositional-defiant, conduct, and anxiety/depression domains. It also includes 8 performance/impairment items scored 1-5 ("Excellent" to "Problematic"). Higher symptom scores (0-141) indicate greater severity of ADHD-related behaviors, while higher performance scores indicate worse functioning.

OTHER OUTCOMES:
Correlation of Cortical Thickness (MRI) with Change in ANT Conflict Effect | MRI obtained once at baseline.
  Cortical thickness (mm) in prefrontal and cingulo-opercular regions measured with MRI at baseline correlated with change in ANT conflict effect (ms).
Correlation of Cortical Volume (MRI) with Change in ANT Conflict Effect | MRI obtained once at baseline.
  Cortical volume (mm³) in prefrontal and cingulo-opercular regions measured with MRI at baseline correlated with change in ANT conflict effect (ms).
Correlation of Genetic Variant Frequencies with Change in ANT Conflict Effect | Saliva samples collected once at baseline.
  Frequencies of alleles/genotypes for pre-specified single-nucleotide polymorphisms (SNPs) associated with higher ASD risk or symptom severity obtained from saliva DNA and correlated with the change in ANT Conflict Effect

CONTACTS AND LOCATIONS:
Locations (2):
- Kazakhstan (2):
  - Neurolab Plus, Almaty
  - Non-profit joint-stock company "Al-Farabi Kazakh National University", Almaty

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD), including demographics, baseline and outcome measures from the Attention Network Task (ANT), SNAP-IV, Vanderbilt ADHD Diagnostic Parent Rating Scale, WISC-V indices, genetic markers (saliva DNA sequencing results limited to specified polymorphisms), structural MRI volumetric data, fNIRS prefrontal oxygenation measures, EEG during ANT, and TMS stimulation parameters, will be shared.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: De-identified data will be made available within 12 months following publication of the main study results and will remain available for at least 5 years thereafter.
Access Criteria: Data will be accessible to qualified researchers at academic or medical institutions upon submission of a justified request. Each request will be reviewed by the study steering committee. Approved researchers will sign a data use agreement to ensure compliance with ethical standards, including prohibiting any attempt to re-identify participants. Data will be distributed via a secure repository.
URL: https://osf.io/49bwa

REFERENCES:
- [Background] Yen C, Valentine EP, Chiang MC. The Use of Transcranial Magnetic Stimulation in Attention Optimization Research: A Review from Basic Theory to Findings in Attention-Deficit/Hyperactivity Disorder and Depression. Life (Basel). 2024 Feb 29;14(3):329. doi: 10.3390/life14030329. PMID 38541654
- [Background] Weaver L, Rostain AL, Mace W, Akhtar U, Moss E, O'Reardon JP. Transcranial magnetic stimulation (TMS) in the treatment of attention-deficit/hyperactivity disorder in adolescents and young adults: a pilot study. J ECT. 2012 Jun;28(2):98-103. doi: 10.1097/YCT.0b013e31824532c8. PMID 22551775
- [Background] Bussing R, Mason DM, Bell L, Porter P, Garvan C. Adolescent outcomes of childhood attention-deficit/hyperactivity disorder in a diverse community sample. J Am Acad Child Adolesc Psychiatry. 2010 Jun;49(6):595-605. doi: 10.1016/j.jaac.2010.03.006. Epub 2010 May 1. PMID 20494269
- [Background] Poliakova E, Conrad AL, Schieltz KM, O'Brien MJ. Using fNIRS to evaluate ADHD medication effects on neuronal activity: A systematic literature review. Front Neuroimaging. 2023;2:1083036. doi: 10.3389/fnimg.2023.1083036. Epub 2023 Jan 24. PMID 37033327
- [Background] Lundervold AJ, Adolfsdottir S, Halleland H, Halmoy A, Plessen K, Haavik J. Attention Network Test in adults with ADHD--the impact of affective fluctuations. Behav Brain Funct. 2011 Jul 27;7:27. doi: 10.1186/1744-9081-7-27. PMID 21794128
- [Background] Le HT, Honma K, Annaka H, Shunxiang S, Murakami T, Hiraoka T, Nomura T. Effectiveness of Transcranial Magnetic Stimulation on Executive Function, Attention, and Memory in Stroke Patients: A Systematic Review and Meta-Analysis. Cureus. 2024 Dec 6;16(12):e75194. doi: 10.7759/cureus.75194. eCollection 2024 Dec. PMID 39759598
- [Background] Hall CL, Guo B, Valentine AZ, Groom MJ, Daley D, Sayal K, Hollis C. The Validity of the SNAP-IV in Children Displaying ADHD Symptoms. Assessment. 2020 Sep;27(6):1258-1271. doi: 10.1177/1073191119842255. Epub 2019 Apr 16. PMID 30991820
- [Background] Fu B, Zhou X, Zhou X, Li X, Chen Z, Zhang Y, Du Q. Efficacy and Safety of Transcranial Magnetic Stimulation for Attention-Deficit Hyperactivity Disorder: A Systematic Review and Meta-Analysis. Brain Behav. 2025 Jan;15(1):e70246. doi: 10.1002/brb3.70246. PMID 39829146
- [Background] Mihalache D, Mazilu D, Crasovan LC. Linear stability analysis of walking vector solitons. Phys Rev E Stat Phys Plasmas Fluids Relat Interdiscip Topics. 1999 Dec;60(6 Pt B):7504-10. doi: 10.1103/physreve.60.7504. PMID 11970700
- [Background] Cools R, D'Esposito M. Inverted-U-shaped dopamine actions on human working memory and cognitive control. Biol Psychiatry. 2011 Jun 15;69(12):e113-25. doi: 10.1016/j.biopsych.2011.03.028. Epub 2011 May 4. PMID 21531388
- [Background] Cho SS, Ko JH, Pellecchia G, Van Eimeren T, Cilia R, Strafella AP. Continuous theta burst stimulation of right dorsolateral prefrontal cortex induces changes in impulsivity level. Brain Stimul. 2010 Jul;3(3):170-6. doi: 10.1016/j.brs.2009.10.002. Epub 2009 Oct 31. PMID 20633446
- [Background] Chen YH, Liang SC, Sun CK, Cheng YS, Tzang RF, Chiu HJ, Wang MY, Cheng YC, Hung KC. A meta-analysis on the therapeutic efficacy of repetitive transcranial magnetic stimulation for cognitive functions in attention-deficit/hyperactivity disorders. BMC Psychiatry. 2023 Oct 17;23(1):756. doi: 10.1186/s12888-023-05261-2. PMID 37845676
- [Background] Chen SY, Tsou MH, Chen KY, Liu YC, Lin MT. Impact of repetitive transcranial magnetic stimulation on cortical activity: a systematic review and meta-analysis utilizing functional near-infrared spectroscopy evaluation. J Neuroeng Rehabil. 2024 Jun 24;21(1):108. doi: 10.1186/s12984-024-01407-9. PMID 38915003
- [Background] Bidwell LC, Gray JC, Weafer J, Palmer AA, de Wit H, MacKillop J. Genetic influences on ADHD symptom dimensions: Examination of a priori candidates, gene-based tests, genome-wide variation, and SNP heritability. Am J Med Genet B Neuropsychiatr Genet. 2017 Jun;174(4):458-466. doi: 10.1002/ajmg.b.32535. PMID 28512748
- [Background] Barth B, Rohe T, Deppermann S, Fallgatter AJ, Ehlis AC. Neural oscillatory responses to performance monitoring differ between high- and low-impulsive individuals, but are unaffected by TMS. Hum Brain Mapp. 2021 Jun 1;42(8):2416-2433. doi: 10.1002/hbm.25376. Epub 2021 Feb 19. PMID 33605509
- [Background] Anderson NP, Feldman JA, Kolko DJ, Pilkonis PA, Lindhiem O. National Norms for the Vanderbilt ADHD Diagnostic Parent Rating Scale in Children. J Pediatr Psychol. 2022 Jun 7;47(6):652-661. doi: 10.1093/jpepsy/jsab132. PMID 34986222
- [Background] Dos Santos Afonso Junior A, Machado-Pinheiro W, Osorio AAC, Seabra AG, Teixeira MCTV, de Araujo Nascimento J, Carreiro LRR. Association between ADHD symptoms and inhibition-related brain activity using functional near-infrared spectroscopy (fNIRS). Neurosci Lett. 2023 Jan 1;792:136962. doi: 10.1016/j.neulet.2022.136962. Epub 2022 Nov 11. PMID 36375626